CLINICAL TRIAL: NCT03729518
Title: A Phase II Study of Volume and Dose De-Intensification Following Transoral Robotic Surgery (TORS) and Neck Dissection for p16+ Oropharyngeal Squamous Cell Carcinoma
Brief Title: TORS De-Intensification Protocol Version 2.0: Dose and Volume Reduction in the Neck
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 15318
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Oropharyngeal Cancer; Squamous Cell Carcinoma; Human Papilloma Virus
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma, Squamous Cell | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Arm 1 (Experimental): All patients will have the volume treated and radiation dose delivered to the regional lymphatics decreased according to the characteristics of the primary site and involved lymph nodes. The high risk neck will receive 50 Gy instead of 60 Gy, and the treated volume of the contralateral low risk neck will be reduced and receive only 45 Gy.
  Interventions: Radiation: Radiation Therapy (IMRT or IMPT)

INTERVENTIONS:
Radiation: Radiation Therapy (IMRT or IMPT) — * Treatment of the primary tumor bed will be omitted in appropriate patients, as per the initial TORS de-intensification protocol. In those patients requiring treatment of the primary site, reduced dose (50 Gy) will be delivered.
  * Receipt of concurrent chemotherapy per current guidelines. Chemotherapy may be omitted in patients with focal or microscopic ENE (defined as ≤ 1 mm ENE), at the discretion of the treating Medical Oncologist.
  * Blood samples will be obtained at time of enrollment, and at two time points during RT, to quantify circulating HPV DNA and perform immune profiling.

SUMMARY:
This is a single-arm Phase II study of adjuvant radiation for locally advanced p16+ oropharyngeal squamous cell carcinoma. The main purpose of this research is to determine the likelihood of cancer growing back in the throat or in the neck two years after completion of radiation if lower doses of radiation are used to a smaller area of the head and neck region than is currently used in standard of care.

DETAILED DESCRIPTION:
This is a single arm Phase II study of adjuvant radiation for locally-advanced p16+ oropharyngeal squamous cell carcinoma. Patients with pT0-T3, N0-N2b, M0 disease (per AJCC 7th ed) with <5 positive lymph nodes, will be eligible. Patients will have undergone TORS primary site resection and ipsilateral neck dissection. Patients will undergo radiation dose reduction and target volume reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old
* Histologically confirmed diagnosis of squamous cell carcinoma of the oropharynx, p16-positive on immunohistochemistry
* Pathologic T0 (unknown primary), T1, T2, or T3 disease (per AJCC 7th Ed)
* Pathologic N0, N1, N2a, or N2b disease (per AJCC 7th Ed), with < 5 positive lymph nodes
* ECOG Performance Status 0-1

Exclusion Criteria:

* Prior radiation therapy to the head and neck
* Presence of T4 disease
* Presence of N2c or N3 neck disease (per AJCC 7th Ed)
* >= 5 lymph nodes
* Presence of distant metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year locoregional control | 2 years
  Number of patients with 2-year locoregional control, defined as control at the primary site and in the neck, in patients undergoing de-intensified radiation to the primary site and regional lymphatics after Transoral Robotic Surgery (TORS) and neck dissection for p16+ oropharyngeal squamous cell carcinoma (OPSCC)

SECONDARY OUTCOMES:
Treatment-related toxicity | 2 years
  Number of participants with treatment-related toxicity as gauged by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. the CTCAE v.5 utilizes a five point scale to report Adverse Events (AEs), defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of medical treatment or procedure that may or may not be considered related to the medical treatment or procedure (cancer.gov)
2-year progression-free survival | 3 years
  Number of participants with 2-year progression-free survival, defined as the length of time during and after treatment that a patient lives with the disease but it does not get worse (nih.gov)
Differences in toxicity between Intensity-modulated radiation therapy (IMRT) and Intensity Modulated Proton Therapy (IMPT) | 1 year
  Differences in toxicity outcomes in patients treated with IMRT versus proton therapy
Number of participants with change in circulating human papillomavirus(HPV) DNA over the course of treatment | 2 years
  Number of patients with a change in circulating HPV cells during the course of treatment, determined using a next generation sequencing (NGS) assay developed to detect HPV DNA in HPV+ oropharyngeal squamous cell carcinoma patients.
Metastasis-free survival | 3 years
  Number of participants with metastasis-free survival
Patient reported quality of life outcomes | 2.5 years
  Patient reported quality of life (QOL) outcomes using MD Anderson Symptom Inventory (MDASI) Head and Neck survey between patients treated with IMRT and IMPT. The MDASI-HN assesses the severity of symptoms in the last 24 hours using a 0-10 scale, with 0 being "not present" and 10 being "as bad as you can imagine". The interference of symptoms in the last 24 hours is assessed using a 0-10 scale, with 0 being "did not interfere" and 10 being "interfered completely". The mean of symptom severity and interference can be used to represent overall symptom distress and can be analyzed for changes over treatment and during follow-up.
Overall survival | 5 years
  Number of patients with overall survival, as defined by the length of time from the date of diagnosis or start of treatment for a disease that patients diagnosed with the disease are still alive (cancer.gov)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinstein GS, O'Malley BW Jr, Cohen MA, Quon H. Transoral robotic surgery for advanced oropharyngeal carcinoma. Arch Otolaryngol Head Neck Surg. 2010 Nov;136(11):1079-85. doi: 10.1001/archoto.2010.191. PMID 21079160
- [Background] Weinstein GS, Quon H, O'Malley BW Jr, Kim GG, Cohen MA. Selective neck dissection and deintensified postoperative radiation and chemotherapy for oropharyngeal cancer: a subset analysis of the University of Pennsylvania transoral robotic surgery trial. Laryngoscope. 2010 Sep;120(9):1749-55. doi: 10.1002/lary.21021. PMID 20717944
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] O'Sullivan B, Huang SH, Siu LL, Waldron J, Zhao H, Perez-Ordonez B, Weinreb I, Kim J, Ringash J, Bayley A, Dawson LA, Hope A, Cho J, Irish J, Gilbert R, Gullane P, Hui A, Liu FF, Chen E, Xu W. Deintensification candidate subgroups in human papillomavirus-related oropharyngeal cancer according to minimal risk of distant metastasis. J Clin Oncol. 2013 Feb 10;31(5):543-50. doi: 10.1200/JCO.2012.44.0164. Epub 2013 Jan 7. PMID 23295795
- [Background] Cohen MA, Weinstein GS, O'Malley BW Jr, Feldman M, Quon H. Transoral robotic surgery and human papillomavirus status: Oncologic results. Head Neck. 2011 Apr;33(4):573-80. doi: 10.1002/hed.21500. Epub 2010 Dec 6. PMID 21425382
- [Background] Quon H, Cohen MA, Montone KT, Ziober AF, Wang LP, Weinstein GS, O'Malley BW Jr. Transoral robotic surgery and adjuvant therapy for oropharyngeal carcinomas and the influence of p16 INK4a on treatment outcomes. Laryngoscope. 2013 Mar;123(3):635-40. doi: 10.1002/lary.22172. Epub 2013 Feb 1. PMID 22588642
- [Background] Ingle CJ, Yip K, Caskie V, Dyson C, Ford A, Scrase CD. Intensity modulated radiotherapy (IMRT) in the management of locally advanced oropharyngeal squamous cell carcinomata (SCC): disease control and functional outcome using the therapy outcome measure (TOM) score--report from a single U.K. institution. Head Neck Oncol. 2010 Oct 14;2:28. doi: 10.1186/1758-3284-2-28. PMID 20946673
- [Background] Lukens JN, Lin A, Gamerman V, Mitra N, Grover S, McMenamin EM, Weinstein GS, O'Malley BW Jr, Cohen RB, Orisamolu A, Ahn PH, Quon H. Late consequential surgical bed soft tissue necrosis in advanced oropharyngeal squamous cell carcinomas treated with transoral robotic surgery and postoperative radiation therapy. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):981-988. doi: 10.1016/j.ijrobp.2014.04.024. Epub 2014 Jun 10. PMID 24928257
- [Background] Weinstein GS, Quon H, Newman HJ, Chalian JA, Malloy K, Lin A, Desai A, Livolsi VA, Montone KT, Cohen KR, O'Malley BW. Transoral robotic surgery alone for oropharyngeal cancer: an analysis of local control. Arch Otolaryngol Head Neck Surg. 2012 Jul;138(7):628-34. doi: 10.1001/archoto.2012.1166. PMID 22801885
- [Background] Ojerholm E, Lukens JN, Ahn PH, Geiger G, Swisher-McClure S, Newman J, Chalian A, Weinstein G, O'Malley BW Jr, Cohen R, Lin A. Benefits of omitting primary site radiation therapy after transoral robotic surgery: Only time will tell. Pract Radiat Oncol. 2017 May-Jun;7(3):e157-e158. doi: 10.1016/j.prro.2016.10.019. Epub 2016 Nov 4. No abstract available. PMID 28094210
- [Background] Gamez ME, Halyard MY, Hinni ML, Hayden RE, Nagel TH, Vargas CE, Wong WW, Curtis KK, Zarka MA, Ma D, Patel SH. Mucosal Sparing Radiation Therapy in Resected Oropharyngeal Cancer. Ann Otol Rhinol Laryngol. 2017 Mar;126(3):185-191. doi: 10.1177/0003489416681580. Epub 2017 Jan 5. PMID 28056518
- [Background] Erratum to: Routman DM, Funk RK, Tangsriwong K, et al. Relapse rates with surgery alone in human papillomavirus-related intermediate- and high-risk group oropharynx squamous cell cancer: A multi-institutional review. Int J Radiat Oncol Biol Phys 2017;99:938-946. Int J Radiat Oncol Biol Phys. 2018 Apr 1;100(5):1304. doi: 10.1016/j.ijrobp.2017.12.286. No abstract available. PMID 29722676
- [Background] ClinicalTrials.gov. Post-operative Adjuvant Treatment for HPV-positive Tumours (PATHOS).
- [Background] Chen AM, Felix C, Wang PC, Hsu S, Basehart V, Garst J, Beron P, Wong D, Rosove MH, Rao S, Melanson H, Kim E, Palmer D, Qi L, Kelly K, Steinberg ML, Kupelian PA, Daly ME. Reduced-dose radiotherapy for human papillomavirus-associated squamous-cell carcinoma of the oropharynx: a single-arm, phase 2 study. Lancet Oncol. 2017 Jun;18(6):803-811. doi: 10.1016/S1470-2045(17)30246-2. Epub 2017 Apr 20. PMID 28434660
- [Background] Huang SH, Waldron J, Bratman SV, Su J, Kim J, Bayley A, Cho J, Giuliani M, Hope A, Ringash J, Hansen A, de Almeida JR, Goldstein D, Perez-Ordonez B, Weinreb I, Tong L, Xu W, O'Sullivan B. Re-evaluation of Ipsilateral Radiation for T1-T2N0-N2b Tonsil Carcinoma at the Princess Margaret Hospital in the Human Papillomavirus Era, 25 Years Later. Int J Radiat Oncol Biol Phys. 2017 May 1;98(1):159-169. doi: 10.1016/j.ijrobp.2017.01.018. Epub 2017 Jan 9. PMID 28258895
- [Background] Expert Panel on Radiation Oncology--Head & Neck Cancer:; Yeung AR, Garg MK, Lawson J, McDonald MW, Quon H, Ridge JA, Saba N, Salama JK, Smith RV, Yom SS, Beitler JJ; American College of Radiology. ACR Appropriateness Criteria(R) ipsilateral radiation for squamous cell carcinoma of the tonsil. Head Neck. 2012 May;34(5):613-6. doi: 10.1002/hed.21993. Epub 2012 Jan 17. PMID 22250010
- [Background] Liu C, Corry J, Peters L. Letter to the editor regarding ACR Appropriateness Criteria for ipsilateral radiation for squamous cell carcinoma of the tonsil. Head Neck. 2013 Mar;35(3):464. doi: 10.1002/hed.23207. Epub 2013 Feb 5. No abstract available. PMID 23386545
- [Background] Liu C, Dutu G, Peters LJ, Rischin D, Corry J. Tonsillar cancer: the Peter MacCallum experience with unilateral and bilateral irradiation. Head Neck. 2014 Mar;36(3):317-22. doi: 10.1002/hed.23297. Epub 2013 Jun 1. PMID 23729387
- [Background] Hu KS, Mourad WF, Gamez M, Safdieh J, Lin W, Jacobson AS, Persky MS, Urken ML, Culliney B, Li Z, Tran TN, Schantz SP, Chadha J, Harrison LB. Low rates of contralateral neck failure in unilaterally treated oropharyngeal squamous cell carcinoma with prospectively defined criteria of lateralization. Head Neck. 2017 Aug;39(8):1647-1654. doi: 10.1002/hed.24806. Epub 2017 May 5. PMID 28474380
- [Background] J. Gershowitz AD, J.N. Lukens, S.D. Swisher-McClure, G.A. Geiger Jr., A. Lin. Pathologic Risk Factors Associated With Contralateral Neck Disease in Patients with Tonsil Cancer: Implications on Patient Selection for Unilateral Neck Radiation Therapy. International Journal of Radiation Oncology Biology Physics. 2017;99(2):S234.
- [Background] H.B. Musunuru PY, H.C. Ko, T. Kennedy, P.M. Harari, M.E. Witek. Can Elective Neck Radiation Treatment Volumes be Safely Reduced to Diminish Toxicity Profiles for Oropharynx Cancer Patients? International journal of radiation oncology, biology, physics. 2017;99(2 Supplement):E361.
- [Background] Sinha P, Lewis JS Jr, Piccirillo JF, Kallogjeri D, Haughey BH. Extracapsular spread and adjuvant therapy in human papillomavirus-related, p16-positive oropharyngeal carcinoma. Cancer. 2012 Jul 15;118(14):3519-30. doi: 10.1002/cncr.26671. Epub 2011 Nov 15. PMID 22086669
- [Background] Kaczmar JM, Tan KS, Heitjan DF, Lin A, Ahn PH, Newman JG, Rassekh CH, Chalian AA, O'Malley BW Jr, Cohen RB, Weinstein GS. HPV-related oropharyngeal cancer: Risk factors for treatment failure in patients managed with primary transoral robotic surgery. Head Neck. 2016 Jan;38(1):59-65. doi: 10.1002/hed.23850. Epub 2015 Apr 6. PMID 25197014
- [Background] Rwigema JM, Langendijk JA, Paul van der Laan H, Lukens JN, Swisher-McClure SD, Lin A. A Model-Based Approach to Predict Short-Term Toxicity Benefits With Proton Therapy for Oropharyngeal Cancer. Int J Radiat Oncol Biol Phys. 2019 Jul 1;104(3):553-562. doi: 10.1016/j.ijrobp.2018.12.055. Epub 2019 Jan 6. PMID 30625409
- [Background] P. Ahn SS, O. Zhou, J.N. Lukens, A. Lin. A Comparative Quality of Life Cohort of Oropharyngeal Squamous Cell (OPSCC) Patients Treated With Volumetric Modulated Radiation Therapy (VMAT) Versus Proton Pencil Beam Scanning (PBS). International journal of radiation oncology, biology, physics. 2016;93(3 Supp):S71.
- [Background] Lee JY, Garcia-Murillas I, Cutts RJ, De Castro DG, Grove L, Hurley T, Wang F, Nutting C, Newbold K, Harrington K, Turner N, Bhide S. Predicting response to radical (chemo)radiotherapy with circulating HPV DNA in locally advanced head and neck squamous carcinoma. Br J Cancer. 2017 Sep 5;117(6):876-883. doi: 10.1038/bjc.2017.258. Epub 2017 Aug 15. PMID 28809864
- [Background] Masterson L, Lechner M, Loewenbein S, Mohammed H, Davies-Husband C, Fenton T, Sudhoff H, Jani P, Goon P, Sterling J. CD8+ T cell response to human papillomavirus 16 E7 is able to predict survival outcome in oropharyngeal cancer. Eur J Cancer. 2016 Nov;67:141-151. doi: 10.1016/j.ejca.2016.08.012. Epub 2016 Sep 24. PMID 27669501
- [Background] Parikh F, Duluc D, Imai N, Clark A, Misiukiewicz K, Bonomi M, Gupta V, Patsias A, Parides M, Demicco EG, Zhang DY, Kim-Schulze S, Kao J, Gnjatic S, Oh S, Posner MR, Sikora AG. Chemoradiotherapy-induced upregulation of PD-1 antagonizes immunity to HPV-related oropharyngeal cancer. Cancer Res. 2014 Dec 15;74(24):7205-16. doi: 10.1158/0008-5472.CAN-14-1913. Epub 2014 Oct 15. PMID 25320012
- [Background] Huang AC, Postow MA, Orlowski RJ, Mick R, Bengsch B, Manne S, Xu W, Harmon S, Giles JR, Wenz B, Adamow M, Kuk D, Panageas KS, Carrera C, Wong P, Quagliarello F, Wubbenhorst B, D'Andrea K, Pauken KE, Herati RS, Staupe RP, Schenkel JM, McGettigan S, Kothari S, George SM, Vonderheide RH, Amaravadi RK, Karakousis GC, Schuchter LM, Xu X, Nathanson KL, Wolchok JD, Gangadhar TC, Wherry EJ. T-cell invigoration to tumour burden ratio associated with anti-PD-1 response. Nature. 2017 May 4;545(7652):60-65. doi: 10.1038/nature22079. Epub 2017 Apr 10. PMID 28397821
- [Background] Kamphorst AO, Pillai RN, Yang S, Nasti TH, Akondy RS, Wieland A, Sica GL, Yu K, Koenig L, Patel NT, Behera M, Wu H, McCausland M, Chen Z, Zhang C, Khuri FR, Owonikoko TK, Ahmed R, Ramalingam SS. Proliferation of PD-1+ CD8 T cells in peripheral blood after PD-1-targeted therapy in lung cancer patients. Proc Natl Acad Sci U S A. 2017 May 9;114(19):4993-4998. doi: 10.1073/pnas.1705327114. Epub 2017 Apr 26. PMID 28446615
- [Background] Tejeda HA, Green SB, Trimble EL, Ford L, High JL, Ungerleider RS, Friedman MA, Brawley OW. Representation of African-Americans, Hispanics, and whites in National Cancer Institute cancer treatment trials. J Natl Cancer Inst. 1996 Jun 19;88(12):812-6. doi: 10.1093/jnci/88.12.812. PMID 8637047
- [Background] Sikora AG, Toniolo P, DeLacure MD. The changing demographics of head and neck squamous cell carcinoma in the United States. Laryngoscope. 2004 Nov;114(11):1915-23. doi: 10.1097/01.mlg.0000147920.66486.bc. PMID 15510014
- [Background] Society AC. Cancer Facts and Figures 2011. 2011.